CLINICAL TRIAL: NCT00140504
Title: Preventing Adverse Drug Events With PatientSite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Blue Cross Blue Shield (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Saul N. Weingart, MD, PhD, VP for Quality Improvement and Patient Safety, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 05-061; Weingart - K08HS11644
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Adverse Drug Event
Keywords: Adverse drug event; Patient safety; Internet portal; PatientSite; Preventive health; Primary care
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- MedCheck (Experimental): Electronic medication safety queries via PatientSite portal
  Interventions: Other: Medcheck message
- Usual care (No Intervention): No electronic medication safety messages via PatientSite portal

INTERVENTIONS:
Other: Medcheck message — Participants selected at random will receive one email message asking them questions about their prescription which will be forwarded to their physician
  Arms: MedCheck

SUMMARY:
This is a study to better understand the nature and extent of adverse drug events (ADEs), defined as injuries due to prescription medications, in primary care. We will study whether PatientSite (an internet-based communication program for patients and health care providers) can improve clinicians' ability to detect adverse drug events among primary care patients and to mitigate the consequences by sending electronic queries to patients after they receive new medication prescriptions.

DETAILED DESCRIPTION:
* A drug safety module called MedCheck was developed for PatientSite. This allows physicians to query patients automatically 10 days after they receive a new prescription asking them questions about their new prescription. In this study new enhancements will be tested.
* Participants will be assigned at random to the intervention group or control group. The intervention group will receive a single electronic PatientSite message asking them questions about the new prescription which is then forwarded to their physician. The control group will receive a generic message about medication safety.
* To identify adverse drug events, a telephone survey and medical record review will be conducted of patients in the intervention group and controls.
* This study will run for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >18
* Patients that receive a new prescription
* Proficient in spoken and written english

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2003-04; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
To prevent adverse drug events with PatientSite. | 3 years

SECONDARY OUTCOMES:
Improve patient satisfaction | 3 years
better utilization of services | 3 years
improve patient-clinician communication | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Saul N Weingart, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Weingart SN, Carbo A, Tess A, Chiappetta L, Tutkus S, Morway L, Toth M, Davis RB, Phillips RS, Bates DW. Using a patient internet portal to prevent adverse drug events: a randomized, controlled trial. J Patient Saf. 2013 Sep;9(3):169-75. doi: 10.1097/PTS.0b013e31829e4b95. PMID 23965840